CLINICAL TRIAL: NCT01296529
Title: A Pilot Study on Immunopathogenesis in HIV and Hepatitis C Coinfection
Brief Title: Study on Immunopathogenesis in HIV and Hepatitis C Coinfection
Status: Completed | Type: Observational
Sponsor: Rush University Medical Center (Other)
Collaborators: Ruth M. Rothstein CORE Center (Other); Merck Sharp & Dohme LLC (Industry); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Gregory Huhn, MD, Rush University Medical Center
Other Study IDs: 100517002
Record Dates: First submitted 2011-01-26; First posted 2011-02-15 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infection; Hepatitis C Infection; Fibrosis; Inflammation
MeSH Terms: conditions — HIV Infections; Hepatitis C; Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- HIV monoinfection: Evidence should include a copy of a laboratory report of testing positive for HIV antibodies and/or HIV viral RNA, and a negative antibody test for HCV
- HCV monoinfection: Evidence should include a copy of a laboratory report of testing positive for HCV antibodies and HCV viral RNA, and a negative antibody test for HIV
- HIV and HCV coinfection: Evidence should include a copy of a laboratory report of testing positive for HIV or HIV viral RNA, and positive tests for HCV antibodies and HCV RNA.
- HIV/HCV coinfection with HCV clearance: Evidence should include a copy of a laboratory report of testing positive for HIV or HIV viral RNA, a positive tests for HCV antibodies, and undetectable HCV RNA without hepatitis C treatment (spontaneous clearance) or >6 months after hepatitis therapy (sustained virologic response)

SUMMARY:
Liver-related death is the leading cause of mortality in HIV-infected individuals with CD4+ cell counts over 200, and hepatitis C virus (HCV) infection is the greatest risk for liver-related mortality in HIV-positive patients. Compared to HCV monoinfected individuals, patients with HIV and HCV coinfection experience accelerated progression of liver fibrosis, which can lead to higher incidence of cirrhosis, end stage liver disease (ESLD), and death. Changes in CD8+ T-cell activation, inflammatory cytokines, and serum markers of tissue injury may offer an immunologic platform to determine factors associated with progressive liver fibrosis in coinfected patients. In this cross-sectional study we will evaluate whether HIV and HCV coinfection patients with well-controlled HIV infection who have an undetectable viral load exhibit abnormal levels of inflammation and immune activation, potentially contributing to advanced liver fibrosis. Comparative groups include coinfected patients successfully treated for hepatitis C, or who have absence of hepatitis C viremia through spontaneous clearance, hepatitis C monoinfected patients, and HIV-positive patients with well-controlled HIV infection without hepatitis C. Liver fibrosis will be measured by non-invasive methods.

The primary objectives of this study are:

1. To determine if there are differences in markers of inflammation and immune activation in subsets of patients with HIV, hepatitis C, and HIV and hepatitis C coinfection.
2. To assess the stage of liver fibrosis using non-invasive methods in subsets of patients with hepatitis C and HIV and hepatitis C coinfection and compare the degree of liver fibrosis with levels of inflammation and immune activation.

ELIGIBILITY:
Inclusion Criteria:

* Strata a (n=15): Patients must be infected with HIV-1 infection without HCV. Evidence should include a copy of a laboratory report of testing positive for HIV antibodies and/or HIV viral RNA, and a negative antibody test for HCV
* Strata b (n=15): Patients must be infected with HCV infection without HIV. Evidence should include a copy of a laboratory report of testing positive for HCV antibodies and HCV viral RNA, and a negative antibody test for HIV
* Strata c (n=15): Patients must be co-infected with HIV & HCV prior to enrollment. Evidence should include a copy of a laboratory report of testing positive for HIV or HIV viral RNA, and positive tests for HCV antibodies and HCV RNA.
* Strata d (n=15): Patients must be co-infected with HIV & HCV prior to enrollment, with verification of successful treatment or spontaneous clearance for hepatitis C infection. Evidence should include a copy of a laboratory report of testing positive for HIV or HIV viral RNA, a positive tests for HCV antibodies, and undetectable HCV RNA without hepatitis C treatment (spontaneous clearance) or >6 months after hepatitis therapy (sustained virologic response)
* Patients should not have ESLD and/or HCC within 6 months of enrollment. Evidence should at least include a physical examination by certified medical practitioner, negative ultrasound of the liver, and laboratory testing consistent with Child A and a Model for ESLD (MELD) ≤ 10. (Note: patients taking atazanavir may be enrolled with elevated total bilirubin if other Child and MELD criteria are normal.)
* Treatment with antiretroviral drugs for at least 12 months
* Undetectable HIV-1 RNA (<75 copies for at least 6 months)
* Patients must consent to study procedures
* Patients must be >18 years of age

Exclusion Criteria:

* Pregnancy
* History of End Stage Liver Disease
* Active hepatitis B infection
* Severe illness / discretion of investigator
* BMI ≥ 35

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: a) HIV monoinfected; b) hepatitis C monoinfected; c) HIV/HCV coinfected untreated for hepatitis C; and d) HIV/HCV coinfected with clearance of HCV virus. Subjects will be all matched by age and estimated duration of hepatitis C infection where applicable. In addition, subjects in strata a and c will be matched by length of ARV therapy and CD4 count first established in strata d observed immediately before the initiation of successful hepatitis C therapy or documentation of negative HCV RNA in subjects with spontaneous clearance. Subjects in strata b will be matched in the same manner to strata d, except length of ARV therapy and CD4 count variables will not be considered. All subjects with HIV infection will be on HAART with undetectable viral loads.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Comparison of liver fibrosis with levels of inflammation and immune activation in subsets of patients with HIV, hepatitis C, and HIV and hepatitis C coinfection | 6 months
  Assess the associations between liver fibrosis as the dependent variable measured as a fibrosis score in kPa with predictor variables (markers of inflammation [IL-1β, IL-6, IL-8, IL10, IL-12, IL-15, IL-17, IL-21, IP10, IFN-γ, TNF-α, macrophage inflammatory protein 1 alpha (CCR7), hsCRP], immune activation and senescence [CD3, CD4, CD8, HLA DR, CD38, Ki67 CD45RA, CCR7, CD28, CD57], and tissue injury [tissue factor]) for groups b, c, and d separately by using linear regression models. Group a is the control arm for the dependent variable.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Huhn, MD, MPHTM, Principal Investigator — The Ruth M. Rothstein CORE Center
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Ruth M. Rothstein CORE Center, Chicago, Illinois

REFERENCES:
- [Result] Hodowanec A, Brady KE, Gao W, Kincaid S, Plants J, Bahk M, Landay A, Huhn G. Differences in CD4+ T-cell Immune Activation in HIV, Hepatitis C (HCV), and HIV/HCV Coinfection Are Influenced by HIV and HCV Infection Status. Abstract MOPE011. 19th International AIDS Conference, Washington DC, July 23, 2012